CLINICAL TRIAL: NCT06846164
Title: Effects of Progressive Resistance Exercises on Range of Motion & Strength and Function Among Athletes With Hamstring Deficit After ACL Reconstruction
Brief Title: Effects of Progressive Resistance Exercises Among Athletes With Hamstring Deficit After ACL Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0409
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy
Keywords: Anterior Cruciate Ligament; resistance training; Athletes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised progressive strength training with elements like (SNG) (Experimental): Participants will be randomized to SNG and perform training sessions (60-70 minutes) twice weekly, over 12 weeks, commencing 8 exercises for the lower extremities in 3 sets of 10 repetitions with an intensity of 12 repetitions maximum. Individual progression, quality of exercise, number of sets, repetitions, and additional training weights will be monitored and adjusted throughout the intervention period by experienced physiotherapists
  Interventions: Other: Supervised progressive strength training including elements of neuromuscular exercise intervention (SNG)
- home based low-intensity weight-bearing exercise protocol (Experimental): Participants allocated to CON will receive written and verbal instructions regarding 4 home-based (low-intensity), weight-bearing exercises for the lower extremities, to be performed twice weekly. This intervention is designed to resemble usual care in cases where persistent knee muscle strength deficits would be discovered and considered a clinical issue.
  Interventions: Other: home based low-intensity weight-bearing exercise protocol.

INTERVENTIONS:
Other: Supervised progressive strength training including elements of neuromuscular exercise intervention (SNG) — Participants will be randomized to SNG and will perform training sessions (60-70 minutes) twice weekly, over a duration of 12 weeks, commencing 8 exercises for the lower extremities in 3 sets of 10 repetitions with an intensity of 12 repetitions maximum. Individual progression, quality of exercise, number of sets, repetitions, and additional training weights will be monitored
  Arms: Supervised progressive strength training with elements like (SNG)
Other: home based low-intensity weight-bearing exercise protocol. — Participants allocated to CON will receive written and verbal instructions regarding 4 home-based (low intensity), weight-bearing exercises for the lower extremities, to be performed twice weekly. This intervention is designed to resemble usual care in cases where persistent knee muscle strength deficits would be discovered and considered a clinical issue.
  Arms: home based low-intensity weight-bearing exercise protocol

SUMMARY:
The goal of the study is to find out how mild home exercises (similar to usual care) and progressive strength training, which include neuromuscular exercise, affected knee joint function and HS muscle strength in individuals who has persistent HS muscle strength deficits 12-24 months after ACLR.

DETAILED DESCRIPTION:
The objective of the present study is to investigate whether individuals, who perform supervised progressive strength training including elements of neuromuscular exercise intervention (SNG) will achieve greater improvements in leg muscle power and greater improvements in knee function compared with individuals performing a homebased low-intensity weight-bearing exercise protocol. We hypothesize that supervised progressive strength training would be superior to a homebased low-intensity weight-bearing exercise protocol for regaining muscle strength and knee function. This study will impact society by promoting health, reducing healthcare costs, supporting productivity, and contributing to a more active and engaged community. Limited investigation exists regarding the durability of progressive resistance exercises in mitigating hamstring deficits post-ACL reconstruction and the personalized optimization of exercise protocols for individual athletes. Further exploration is needed for sustained benefits and tailored rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 30 years
* 12-24 months post-surgery (ACL reconstruction)
* Persistent maximal isometric knee flexor strength asymmetry (>10% leg-to-leg the difference, in the isometric testing angle of 90° knee flexion)

Exclusion Criteria:

* Body mass index [BMI] more than 35
* known lower limb pathology (including previous and/or concomitant knee injuries requiring surgical intervention to either knee)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Limb Symmetry Index | 12 weeks
  It is used for knee extensors and flexors strength. It is the strength ratio between the injured and uninjured knees. It is a common method of assessing strength and functional performance after ACLR.

SECONDARY OUTCOMES:
H/Q ratio | 12 weeks
  it is used to detect muscle imbalance, monitor knee joint stability, and indicate lower extremity injury prevention and rehabilitation.

OTHER OUTCOMES:
KOOS questionnaire | 12 weeks
  It is used to assess five outcomes: pain, activity of daily living, sport and recreation function, and knee-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Attiq ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Innovative Health Concept, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chechik O, Amar E, Khashan M, Lador R, Eyal G, Gold A. An international survey on anterior cruciate ligament reconstruction practices. Int Orthop. 2013 Feb;37(2):201-6. doi: 10.1007/s00264-012-1611-9. Epub 2012 Jul 11. PMID 22782378
- [Background] Mall NA, Chalmers PN, Moric M, Tanaka MJ, Cole BJ, Bach BR Jr, Paletta GA Jr. Incidence and trends of anterior cruciate ligament reconstruction in the United States. Am J Sports Med. 2014 Oct;42(10):2363-70. doi: 10.1177/0363546514542796. Epub 2014 Aug 1. PMID 25086064
- [Background] Shaerf DA, Pastides PS, Sarraf KM, Willis-Owen CA. Anterior cruciate ligament reconstruction best practice: A review of graft choice. World J Orthop. 2014 Jan 18;5(1):23-9. doi: 10.5312/wjo.v5.i1.23. eCollection 2014 Jan 18. PMID 24649411
- [Background] Ardern CL, Webster KE, Taylor NF, Feller JA. Return to the preinjury level of competitive sport after anterior cruciate ligament reconstruction surgery: two-thirds of patients have not returned by 12 months after surgery. Am J Sports Med. 2011 Mar;39(3):538-43. doi: 10.1177/0363546510384798. Epub 2010 Nov 23. PMID 21098818
- [Background] Filbay SR, Grindem H. Evidence-based recommendations for the management of anterior cruciate ligament (ACL) rupture. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):33-47. doi: 10.1016/j.berh.2019.01.018. Epub 2019 Feb 21. PMID 31431274
- [Background] Gobbi A, Francisco R. Factors affecting return to sports after anterior cruciate ligament reconstruction with patellar tendon and hamstring graft: a prospective clinical investigation. Knee Surg Sports Traumatol Arthrosc. 2006 Oct;14(10):1021-8. doi: 10.1007/s00167-006-0050-9. Epub 2006 Feb 22. PMID 16496124
- [Background] Bram JT, Magee LC, Mehta NN, Patel NM, Ganley TJ. Anterior Cruciate Ligament Injury Incidence in Adolescent Athletes: A Systematic Review and Meta-analysis. Am J Sports Med. 2021 Jun;49(7):1962-1972. doi: 10.1177/0363546520959619. Epub 2020 Oct 22. PMID 33090889
- [Background] Bencke J, Aagaard P, Zebis MK. Muscle Activation During ACL Injury Risk Movements in Young Female Athletes: A Narrative Review. Front Physiol. 2018 May 15;9:445. doi: 10.3389/fphys.2018.00445. eCollection 2018. PMID 29867521
- [Background] More RC, Karras BT, Neiman R, Fritschy D, Woo SL, Daniel DM. Hamstrings--an anterior cruciate ligament protagonist. An in vitro study. Am J Sports Med. 1993 Mar-Apr;21(2):231-7. doi: 10.1177/036354659302100212. PMID 8465918
- [Background] Zebis MK, Andersen LL, Bencke J, Kjaer M, Aagaard P. Identification of athletes at future risk of anterior cruciate ligament ruptures by neuromuscular screening. Am J Sports Med. 2009 Oct;37(10):1967-73. doi: 10.1177/0363546509335000. Epub 2009 Jul 2. PMID 19574475
- [Background] Bieler T, Sobol NA, Andersen LL, Kiel P, Lofholm P, Aagaard P, Magnusson SP, Krogsgaard MR, Beyer N. The effects of high-intensity versus low-intensity resistance training on leg extensor power and recovery of knee function after ACL-reconstruction. Biomed Res Int. 2014;2014:278512. doi: 10.1155/2014/278512. Epub 2014 Apr 27. PMID 24877078
- [Background] Hanada M, Yoshikura T, Matsuyama Y. Muscle recovery at 1 year after the anterior cruciate ligament reconstruction surgery is associated with preoperative and early postoperative muscular strength of the knee extension. Eur J Orthop Surg Traumatol. 2019 Dec;29(8):1759-1764. doi: 10.1007/s00590-019-02479-3. Epub 2019 Jun 25. PMID 31240385